CLINICAL TRIAL: NCT05656768
Title: Sleep and Circadian Contributions to Nighttime Blood Pressure
Acronym: SCN-BP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stephen Justin Thomas, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300010042
Record Dates: First submitted 2022-11-18; First posted 2022-12-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Circadian Rhythm; Blood Pressure; Hypertension
Keywords: sleep; circadian rhythm; circadian misalignment; nocturnal hypertension; non-dipping blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Constant Routine Protocol (Experimental): Participants complete a 30-hour constant routine protocol to directly examine markers of endogenous circadian rhythms. In a constant routine protocol, participants remain in a dimly lit room (<10 lux), in a semi-recumbent posture, remain awake, and consume iso-caloric snacks. Saliva samples are collected and core body temperature and blood pressure are measured.
  Interventions: Other: Constant Routine Protocol

INTERVENTIONS:
Other: Constant Routine Protocol — A constant routine protocol is used to directly examine markers of circadian rhythmicity (e.g., melatonin and core body temperature). A constant routine protocol requires an individual to remain in a dimly lit room, in a constant semi-recumbent posture, and remain awake for more than 24 hours. It is one of two gold-standard research protocols for examining circadian rhythms in humans.

SUMMARY:
Broadly, this study (SCN-BP) seeks to examine sleep and circadian factors that contribute to blood pressure levels at night.

DETAILED DESCRIPTION:
SCN-BP is imbedded in a parent grant titled "Improving the Detection of Hypertension (IDH-MEGA)" and examines a variety of sleep (e.g., sleep duration, timing, and the presence of sleep disorder) and circadian factors in Aims 1 and 2. In Aim 3, the investigators will conduct a 30-hour constant routine protocol to directly examine endogenous circadian and blood pressure rhythms. Aims 1 and 2 are purely observation. The study design design described below pertains the intervention piece of this study (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Participant in the parent grant (IDH-MEGA)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1427 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Melatonin | Hourly samples obtained over 30 hours
  Melatonin levels obtained from saliva samples
Change in Core body temperature | Continuous measurements over 30 hours
  Core body temperature

SECONDARY OUTCOMES:
Change in Blood pressure | Measurements obtained every 30 minutes over 30 hours
  Systolic and diastolic blood pressure obtained using an ambulatory blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Thomas, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States